CLINICAL TRIAL: NCT02381249
Title: The Effect of Satiety Gut Hormone Modulation on Appetitive Drive After Upper Gastrointestinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: University College Dublin (Other); University of Dublin, Trinity College (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRFSJ 0057
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition; Pancreatic Neoplasms; Duodenal Neoplasms
Keywords: Esophagectomy; Gastrectomy; Octreotide; Somatostatin; Appetite; Hunger; Glucagon-Like Peptide 1; Peptide YY; Reinforcement; Reward; Psychological Phenomena and Processes; Gastrointestinal Agents; Nutritional Status; Pancreaticoduodenectomy; Whipple Procedure
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Weight Loss; Malnutrition; Pancreatic Neoplasms; Duodenal Neoplasms | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Esophagectomy (Experimental): Double-blind single dose octreotide-placebo crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Gastrectomy (Experimental): Double-blind single dose octreotide-placebo crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Unoperated healthy control (Active Comparator): Double-blind single dose octreotide-placebo crossover
  Interventions: Drug: Octreotide; Drug: Placebo
- Pancreaticoduodenectomy (Experimental): Double-blind single dose octreotide-placebo crossover
  Interventions: Drug: Octreotide; Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Single dose 100mcg octreotide acetate (1mL), subcutaneously to the lower abdomen
  Other Names: Sandostatin
Drug: Placebo — Single dose 0.9% saline (1mL), subcutaneously to the lower abdomen

SUMMARY:
Improvements to treatment strategies for patients with cancers of the upper gastrointestinal tract have produced a large population of people who remain free from cancer recurrence in the long term following treatment.

Surgery is the cornerstone of treatment for patients with these cancers, but while surgical removal of the tumour may offer the best chance of cure, these are major operations associated with specific long term complications. Weight loss and poor nutrition are common problems among patients who attain long-term cancer remission and cure after surgery. The mechanisms underlying these problems are not well understood and therefore treatment options are limited.

Our research has demonstrated increased levels of chemical messengers (gut hormones) released from the gastrointestinal tract after meals in patients who have previously undergone this type of surgery. These chemical messengers play a role in controlling appetite and interest in food, and increased levels after surgery may reduce interest in eating. Understanding the role of gut hormones in the control of appetite may allow us to use certain medications to block gut hormones and hence increase appetite, allowing patients to eat more and regain weight, preventing nutritional problems after surgery.

In this study, the investigators aim to determine whether exaggerated gut hormone secretion causes reduced appetite and interest in food after surgery. The information gained from this study may help us to develop treatments for patients with weight loss and nutritional problems after surgery.

ELIGIBILITY:
Inclusion criteria:

1. Surgical procedure: Two-stage, three-stage or transhiatal esophagectomy with gastric conduit reconstruction and pyloroplasty, total gastrectomy with Roux-en-Y reconstruction, pancreaticoduodenectomy, or matched healthy unoperated control subjects
2. Disease-free at least one year post-resection

Exclusion criteria:

1. Pregnancy, breastfeeding
2. Significant and persistent chemoradiotherapy and/or surgical complication
3. Other previous upper gastrointestinal surgery
4. Unwell or unable to eat
5. Other disease or medications which may affect satiety gut hormone responses
6. Active and significant psychiatric illness including substance misuse
7. Cognitive or communication issues or any factors affecting capacity to consent to participation
8. History of significant food allergy, certain dietary restrictions
9. Confirmed or suspected residual or recurrent disease after surgery, second primary malignancy
10. Requiring adjuvant chemotherapy
11. Contraindication to octreotide administration
12. History of eating disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Progressive ratio task breakpoint for a sweet-fat reward | 3 hours

SECONDARY OUTCOMES:
Number of rewards consumed | 3 hours
Subjective symptom score | 3 hours

OTHER OUTCOMES:
Sigstad score | 3 hours
  Both categorical and continuous

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MCh, FRCS, Principal Investigator — Department of Surgery, St. James's Hospital
Locations (2):
- Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin, Ireland
- Gastrosurgical Laboratory, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Background] Miras AD, Jackson RN, Jackson SN, Goldstone AP, Olbers T, Hackenberg T, Spector AC, le Roux CW. Gastric bypass surgery for obesity decreases the reward value of a sweet-fat stimulus as assessed in a progressive ratio task. Am J Clin Nutr. 2012 Sep;96(3):467-73. doi: 10.3945/ajcn.112.036921. Epub 2012 Jul 25. PMID 22836034
- [Background] HODOS W. Progressive ratio as a measure of reward strength. Science. 1961 Sep 29;134(3483):943-4. doi: 10.1126/science.134.3483.943. PMID 13714876
- [Background] Miholic J, Orskov C, Holst JJ, Kotzerke J, Pichlmayr R. Postprandial release of glucagon-like peptide-1, pancreatic glucagon, and insulin after esophageal resection. Digestion. 1993;54(2):73-8. doi: 10.1159/000201016. PMID 8319842
- [Background] Haverkort EB, Binnekade JM, Busch OR, van Berge Henegouwen MI, de Haan RJ, Gouma DJ. Presence and persistence of nutrition-related symptoms during the first year following esophagectomy with gastric tube reconstruction in clinically disease-free patients. World J Surg. 2010 Dec;34(12):2844-52. doi: 10.1007/s00268-010-0786-8. PMID 20842361
- [Background] Koizumi M, Hosoya Y, Dezaki K, Yada T, Hosoda H, Kangawa K, Nagai H, Lefor AT, Sata N, Yasuda Y. Postoperative weight loss does not resolve after esophagectomy despite normal serum ghrelin levels. Ann Thorac Surg. 2011 Apr;91(4):1032-7. doi: 10.1016/j.athoracsur.2010.11.072. PMID 21440118
- [Background] le Roux CW, Aylwin SJ, Batterham RL, Borg CM, Coyle F, Prasad V, Shurey S, Ghatei MA, Patel AG, Bloom SR. Gut hormone profiles following bariatric surgery favor an anorectic state, facilitate weight loss, and improve metabolic parameters. Ann Surg. 2006 Jan;243(1):108-14. doi: 10.1097/01.sla.0000183349.16877.84. PMID 16371744
- [Derived] Elliott JA, Docherty NG, Haag J, Eckhardt HG, Ravi N, Reynolds JV, le Roux CW. Attenuation of satiety gut hormones increases appetitive behavior after curative esophagectomy for esophageal cancer. Am J Clin Nutr. 2019 Feb 1;109(2):335-344. doi: 10.1093/ajcn/nqy324. PMID 30722001
- See also: Wellcome Trust-HRB Clinical Research Facility — http://www.sjhcrf.ie